CLINICAL TRIAL: NCT00116987
Title: Pacing the Octogenarian Plus Population (POPP) A Comparison of Physiologic Versus Ventricular Pacing in Those Who Are 80 Years of Age and Older
Brief Title: Dual Chamber Versus Single Chamber Cardiac Pacing in People 80 Years of Age and Older
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit adequate number of participants in required time frame.
Sponsor: University of Calgary (Other)
Collaborators: Calgary Health Trust (Other)
Responsible Party: Principal Investigator, Dr. Anne M. Gillis, Professor of Medicine, University of Calgary, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17096
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Atrial Fibrillation; Cardiac Pacing, Artificial
Keywords: physiologic pacing; ventricular pacing; hospitalizations
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Physiologic pacemakers usually have two leads - one positioned in the right atrium (upper heart chamber) and one positioned in the right ventricle.
  Interventions: Device: Dual chamber cardiac pacemaker
- 2 (Other): Ventricular pacemakers have a single lead (wire) positioned in the right ventricle (lower pumping chamber) to sense and pace the ventricle.
  Interventions: Device: Single chamber cardiac pacemaker

INTERVENTIONS:
Device: Dual chamber cardiac pacemaker — Physiologic pacemakers usually have two leads - one positioned in the right atrium (upper heart chamber) and one positioned in the right ventricle.
  Arms: 1
Device: Single chamber cardiac pacemaker — Ventricular pacemakers have a single lead (wire) positioned in the right ventricle (lower pumping chamber) to sense and pace the ventricle.
  Arms: 2

SUMMARY:
Of the 19,000 pacemakers implanted across Canada in 2002, 1/3 of them were for patients 80 years and older. This is the fastest growing segment of our population, yet no study has specifically been done in this age group to determine the optimal pacing mode.

We wish to determine whether dual chamber or single chamber pacing is associated with a reduction in emergency room visits or hospitalizations for cardiovascular causes (e.g., congestive heart failure (CHF), atrial fibrillation (AF)) resulting in improved quality of life.

DETAILED DESCRIPTION:
Many patients who are 80 years of age and older, develop AF or CHF. Physiologic pacing has been shown to prevent AF compared to ventricular pacing. Whether prevention of AF and CHF by physiologic pacing reduces emergency room visits or hospitalizations for cardiovascular causes in this population in unknown.

The investigators wish to determine the optimal pacing mode for this patient population that would enable optimal management of cardiovascular problems, resulting in improved quality of life and minimizing use of health care facilities.

Patients recruited to the study will be randomized to either DDDR or VVIR pacing, and followed in the clinic every 6 months for the 3 years of the study.

ELIGIBILITY:
Inclusion Criteria:

* 80 years of age and older
* Symptomatic bradycardia

Exclusion Criteria:

* Permanent atrial fibrillation
* Previous pacemaker implant
* Life expectancy less than 1 year
* Geographic isolation
* Unable to give informed consent

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2003-08; Primary Completion 2008-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To determine which pacing mode, physiologic or ventricular, is associated with a reduction in emergency room visits or hospitalizations for cardiovascular/cerebrovascular causes | approximately 3 - 5 years

SECONDARY OUTCOMES:
To determine which pacing mode, physiologic or ventricular, is associated with improved functional capacity and improved quality of life | approximately 3 - 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Gillis, MD, Principal Investigator — Director of Pacing and Electrophysiology, Professor of Medicine, University of Calgary; Derek V Exner, MD, MPH, Study Director — University of Calgary; D. George Wyse, MD, PhD, Study Director — University of Calgary; L. Brent Mitchell, MD, Study Director — University of Calgary; Robert S Sheldon, MD, Ph D, Study Director — University of Calgary; John M Rothschild, MD, Study Director — University of Calgary; Henry J Duff, MD, Study Director — University of Calgary; John Burgess, MD, Study Director — University of Calgary; Alexander Bayes, MD, Study Director — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada